CLINICAL TRIAL: NCT04677764
Title: Efficacy of Wii Fit Training on Lower Limb Burn in Adults
Brief Title: Virtual Reality in Lower Limb Adult Burn
Acronym: adultburn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, Department of Physical Therapy, College of Medical Rehabilitation, Qassim University, Saudi Arabia, Qassim, Buraidah., Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2657PT
Record Dates: First submitted 2020-12-11; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Burns
Keywords: burns; lower limb burns; virtual reality
MeSH Terms: conditions — Burns | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded author to group allocation collected the outcome measures at baseline and after 12 weeks of intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wii Fit Group (Experimental): Received Standard of care and Wii Fit protocol consisted of strength, balance, and aerobic programs that were performed on the Wii Fit balance board (Nintendo Inc., Kyoto, Japan). For muscle strengthening exercise, lunges, single-leg extensions, sideways leg lifts, single leg twists, and rowing squats were performed. For exercise that enhances balancing sense, the soccer heading, ski slalom, penguin, table tilt, and balance bubble games were used. Aerobic games as hula hoop, super hula hoop and basic step.
  Interventions: Other: virtual reality; Other: Standard of care
- Standard of care group (Other): On discharge from the hospital, patients in the SOC group were given instructions on how to perform physical therapy and occupational therapy exercises after discharge. After education, patients could perform the physical therapy and occupational therapy exercises either at their own home or a gym.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: virtual reality — Wii Fit balance board (Nintendo Inc., Kyoto, Japan).
  Other Names: interactive video games
  Arms: Wii Fit Group
Other: Standard of care — physical therapy and occupational therapy exercises either at their own home or a gym
  Other Names: routine physical therapy protocol

SUMMARY:
To investigate the potential effects of Wii fit rehabilitation programs on functional capacity, mobility, balance and muscle strength in lower limb burn patients after hospital discharge.

DETAILED DESCRIPTION:
The use of virtual reality technology in burn conditions improved joint flexibility and reduced pain associated with physical therapy, dressing changes, and wound debridement. However, the primary concern of burn rehabilitation is not only survival but also maximizing functional outcome and decreasing the time for return to work.

ELIGIBILITY:
Inclusion Criteria:

* adult with a deep partial thickness or a full thickness burn in the lower extremities.
* induced by either a scaled or a flame thermal burn.
* total body surface area (TBSA) more than 40%.
* age ranged from 18 to 40 years.
* recent hospital discharge.

Exclusion Criteria:

* Infection.
* Diabetes.
* inhalation injury.
* Fracture.
* degenerative joint diseases of the lower extremities.
* peripheral nerve diseases.
* Pre-established psychologically and physically disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
high mobility assessment tool | at baseline
  used to assess mobility assessment after burn injuries. It is a valid and reliable unidimensional assessment tool which includes nine functional tasks, where 0 = inability to do and 4= able to do extremely well, with a total score of 54. Each Functional task is rated on a five-point performance scale with higher scores indicate a higher level of performance
high mobility assessment tool | after 12 weeks
  used to assess mobility assessment after burn injuries. It is a valid and reliable unidimensional assessment tool which includes nine functional tasks, where 0 = inability to do and 4= able to do extremely well, with a total score of 54. Each Functional task is rated on a five-point performance scale with higher scores indicate a higher level of performance
Lower Limb Functional Index | at baseline
  a valid and reliable patient self-reported questionnaire to assess lower limb function for patients with a burn injury. It is consisted of fifteen general and ten lower-limb specific items that assess the functional status of the patients during the last 2-3 days. The scoring options for the LLFI Items are Yes=1 point, Somewhat= 0.5 point and No= 0 point. The scoring points are added and then multiplied by four for a total score of functional limitation. The total score of the LLFI ranges from 0 (maximum limitation) to 100 (no limitation or normal functional status)
Lower Limb Functional Index | after 12 weeks
  a valid and reliable patient self-reported questionnaire to assess lower limb function for patients with a burn injury. It is consisted of fifteen general and ten lower-limb specific items that assess the functional status of the patients during the last 2-3 days. The scoring options for the LLFI Items are Yes=1 point, Somewhat= 0.5 point and No= 0 point. The scoring points are added and then multiplied by four for a total score of functional limitation. The total score of the LLFI ranges from 0 (maximum limitation) to 100 (no limitation or normal functional status)
Timed-up and go test | at baseline
  used to evaluate functional mobility of the patients that requires both static and dynamic balance. The TUG test is a basic mobility assessment tool which records the time taken to stand up from a chair, walk 3 meters, return and sit down on the chair. The TUG test was performed with a standardized instruction, asking patients to walk as fast as possible during the test. All participants performed the TUG test from a standard chair (seat height of approximately 46 cm) with back support and no arms
Timed-up and go test | after 12 weeks
  used to evaluate functional mobility of the patients that requires both static and dynamic balance. The TUG test is a basic mobility assessment tool which records the time taken to stand up from a chair, walk 3 meters, return and sit down on the chair. The TUG test was performed with a standardized instruction, asking patients to walk as fast as possible during the test. All participants performed the TUG test from a standard chair (seat height of approximately 46 cm) with back support and no arms

SECONDARY OUTCOMES:
The six-minute walk test | at baseline
  used to assess functional exercise capacity of the participants. The 6-MWT was performed in a 30-meters flat corridor according to the American Thoracic Society guidelines. Patients were asked to walk as far as possible in the 30-m corridor during the 6-min period. Standardized verbal encouragement is given to the patients during the 6-MWT. At the end of the test, the walking distance was measured. The predicted values of 6-MWT were calculated according to age and gender
The six-minute walk test | after 12 weeks
  used to assess functional exercise capacity of the participants. The 6-MWT was performed in a 30-meters flat corridor according to the American Thoracic Society guidelines. Patients were asked to walk as far as possible in the 30-m corridor during the 6-min period. Standardized verbal encouragement is given to the patients during the 6-MWT. At the end of the test, the walking distance was measured. The predicted values of 6-MWT were calculated according to age and gender
Isokinetic Muscle Strength Assessment | at baseline
  assessed by A Biodex dynamometer (Biodex Medical System, Shirley, NY, USA). The values of knee flexors and extensors muscle peak torque of dominant leg were measured regardless the location of burns at an angular velocity of 150°/seconds, hip angle of 100° and patient were supported with a securing belt placed over the mid- thigh, pelvis and trunk. Three sub-maximal repetitions were allowed for the patient without any load as a warm-up. The patient then carried out 10 of maximum voluntary muscle contractions continuously without rest and the highest values were recorded for analysis.
Isokinetic Muscle Strength Assessment | after 12 weeks
  assessed by A Biodex dynamometer (Biodex Medical System, Shirley, NY, USA). The values of knee flexors and extensors muscle peak torque of dominant leg were measured regardless the location of burns at an angular velocity of 150°/seconds, hip angle of 100° and patient were supported with a securing belt placed over the mid- thigh, pelvis and trunk. Three sub-maximal repetitions were allowed for the patient without any load as a warm-up. The patient then carried out 10 of maximum voluntary muscle contractions continuously without rest and the highest values were recorded for analysis.
Stability Index | at baseline
  assessed by A Biodex Balance System (Biodex Medical Systems, Shirley, NY) which consists of a movable balance platform that provides 20° surface tilt through 360° range of motion. The platform interfaces with computer software that enables the device to serve as an objective assessment of balance. All measurements were performed at level eight of stability, and the test duration was set at 20 seconds for three successive trials.
Stability Index | after 12 weeks
  assessed by A Biodex Balance System (Biodex Medical Systems, Shirley, NY) which consists of a movable balance platform that provides 20° surface tilt through 360° range of motion. The platform interfaces with computer software that enables the device to serve as an objective assessment of balance. All measurements were performed at level eight of stability, and the test duration was set at 20 seconds for three successive trials.

CONTACTS AND LOCATIONS:
Overall Officials: Maged Basha, Principal Investigator — Qassim University

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: IPD will be available upon reasonable request by email from the main author after revising the requester qualification relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Result] Jeschke MG, Chinkes DL, Finnerty CC, Kulp G, Suman OE, Norbury WB, Branski LK, Gauglitz GG, Mlcak RP, Herndon DN. Pathophysiologic response to severe burn injury. Ann Surg. 2008 Sep;248(3):387-401. doi: 10.1097/SLA.0b013e3181856241. PMID 18791359
- [Result] Dyster-Aas J, Kildal M, Willebrand M. Return to work and health-related quality of life after burn injury. J Rehabil Med. 2007 Jan;39(1):49-55. doi: 10.2340/16501977-0005. PMID 17225038
- [Result] Kim KJ, Heo M. Effects of virtual reality programs on balance in functional ankle instability. J Phys Ther Sci. 2015 Oct;27(10):3097-101. doi: 10.1589/jpts.27.3097. Epub 2015 Oct 30. PMID 26644652
- [Derived] Basha MA, Abdel-Aal NM, Kamel FAH. Effects of Wii Fit Rehabilitation on Lower Extremity Functional Status in Adults With Severe Burns: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Feb;103(2):289-296. doi: 10.1016/j.apmr.2021.08.020. Epub 2021 Sep 24. PMID 34571011